CLINICAL TRIAL: NCT02443207
Title: Perceived Impact of Dental Pain on the Quality of Life of Preschool Children and Their Families
Brief Title: Impact of Dental Pain on the Quality of Life
Status: Completed | Type: Observational
Sponsor: Ana Flavia Granville-Garcia (Other)
Responsible Party: Sponsor-Investigator, Ana Flavia Granville-Garcia, DDS, PhD, Professor, Universidade Estadual da Paraiba
Organization: Universidade Estadual da Paraiba (Other)
Other Study IDs: CNPq 471-790.2011/7
Record Dates: First submitted 2015-05-06; First posted 2015-05-13 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Dental Pain; Dental Caries
Keywords: Toothache; Quality of life; Oral Health; Children
MeSH Terms: conditions — Toothache; Dental Caries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the present study was to evaluate the perceived impact of dental caries and dental pain on oral health-related quality of life (OHRQoL) among preschool children and their families. A cross-sectional study was conduct with 843 preschool children in Campina Grande, Brazil. Parents/caregivers answered a questionnaire on socio-demographic information, their child's general/oral health and history of dental pain. The Brazilian version of the Early Childhood Oral Health Impact Scale was administered to determine the perceived impact of caries and dental pain on OHRQoL. Children have undergone an oral examination. Logistic regression for complex sample was used to determine associations between the dependent and independent variables (OR: odds ratio; α = 5%).

DETAILED DESCRIPTION:
The present study received approval from the Human Research Ethics Committee of the State University of Paraíba (Brazil) under process number 00460133000-11 in compliance with Resolution 196/96 of the Brazilian National Health Council.

A school-based, cross-sectional study was carried out involving male and female children aged three to five years enrolled at private and public preschools in the city of Campina Grande, Brazil. Campina Grande is an industrialized city in northeastern Brazil with a population of 386,000 inhabitants and is divided into six administrative districts. The city has considerable cultural, social and economic disparities, with a mean monthly income per capita equal to US$ 110 and a Human Development Index of 0.72 [11]. The participants were selected from a total population of 12,705 children in this age group and corresponded to 6.41% of the entire population and therefore representative of preschool children in Campina Grande.

A two-phase sampling method was used to ensure representativeness. A list of preschools was obtained from the Municipal Secretary of Education of Campina Grande. To ensure the representativeness a sample calculation was done. Through a stratified sampling procedure, preschools were selected at draw from each district of Campina Grande. Then the number of schoolchildren from each preschool was proportional to the number of schoolchildren enrolled in each district. The sample was obtained from the proportion estimation calculation. Preschools were randomly selected by draw from each district in the first phase and children were randomly selected from each preschool in the second phase. Eighteen of the 127 public preschools and 15 of the 122 private preschools were randomly selected by lots. The sample size was calculated with a 4% margin of error, a 95% confidence level and a 50% prevalence rate of perceived impact on child and family OHRQoL. A correction factor of 1.2 was applied to compensate for the design effect [12].

The minimum sample size was estimated at 720 schoolchildren, to which an additional 20% was added to compensate for possible losses, giving a total sample of 864 schoolchildren.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were age three to five years of age, enrollment in preschool or daycare and free of any systemic disease according to parents'/caregivers' reports.
* Parental authorization was required and was obtained through a signed statement of informed consent.

Exclusion Criteria:

* Children that did not accept clinical examination or have mental illness were excluded from the study

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A school-based, cross-sectional study was carried out involving male and female children aged three to five years enrolled at private and public preschools in the city of Campina Grande, Brazil. Campina Grande is an industrialized city in northeastern Brazil with a population of 386,000 inhabitants and is divided into six administrative districts. The city has considerable cultural, social and economic disparities, with a mean monthly income per capita equal to US$ 110 and a Human Development Index of 0.72 [11]. The participants were selected from a total population of 12,705 children in this age group and corresponded to 6.41% of the entire population and therefore representative of preschool children in Campina Grande.
Sampling Method: Probability Sample
Enrollment: 843 (Actual)
Dates: Start 2013-01; Primary Completion 2013-09 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Dental Pain | nine months
  Self-reported dental pain informed in a questionnaire
Quality of life | nine months
  Self-reported dental pain informed in a questionnaire (OHRQoL)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Flavia Granville-Garcia, Professor, Principal Investigator — UEPB

REFERENCES:
- [Background] Pahel BT, Rozier RG, Slade GD. Parental perceptions of children's oral health: the Early Childhood Oral Health Impact Scale (ECOHIS). Health Qual Life Outcomes. 2007 Jan 30;5:6. doi: 10.1186/1477-7525-5-6. PMID 17263880
- [Background] Ismail AI, Sohn W, Tellez M, Amaya A, Sen A, Hasson H, Pitts NB. The International Caries Detection and Assessment System (ICDAS): an integrated system for measuring dental caries. Community Dent Oral Epidemiol. 2007 Jun;35(3):170-8. doi: 10.1111/j.1600-0528.2007.00347.x. PMID 17518963
- [Result] Clementino MA, Pinto-Sarmento TC, Costa EM, Martins CC, Granville-Garcia AF, Paiva SM. Association between oral conditions and functional limitations in childhood. J Oral Rehabil. 2015 Jun;42(6):420-9. doi: 10.1111/joor.12273. Epub 2015 Jan 19. PMID 25597878